CLINICAL TRIAL: NCT02318147
Title: Fecal Microbiota Transplantation in SAP（Severe Acute Pancreatitis）Patients With Infectious Complications
Brief Title: Fecal Microbiota Transplantation for Pancreatitis With Infectious Complications(FMTPIC)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lingyu Luo, Physician-in-charge, The First Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NanchanguniversityII
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Acute Pancreatitis; Fecal Microbiota Transplantation; Bacterial Translocation; Infectious Complications
Keywords: Severe acute pancreatitis; Fecal Microbiota Transplantation; Bacterial Translocation; Infectious Complications
MeSH Terms: conditions — Pancreatitis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fecal Microbiota Transplantation (Experimental): FMT by retention enema with fresh bacteria from healthy donor，At the same time give patients the traditional treatment of SAP
  Interventions: Procedure: Fecal Microbiota Transplantation; Drug: The traditional treatment
- The traditional treatment (Other): The traditional treatment of SAP according to the associated guidelines
  Interventions: Drug: The traditional treatment

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — FMT by retention enema with fresh bacteria from healthy donor
  Other Names: Fecal Microbiota Therapy; Fecal Transplantation
  Arms: Fecal Microbiota Transplantation
Drug: The traditional treatment — the traditional treatments according to associated guidelines
  Other Names: Conventional drugs according to the guideline

SUMMARY:
Infectious complications are responsible for most of deaths in acute pancreatitis.Intestinal barrier dysfunction and increased intestinal permeability was associated with bacterial translocation which is believed to prompted these infections.The purpose of this clinical trail is to observe the potential capability of FMT in reduce the bacterial translocation and alleviate infectious complications by the reconstruction of a gut functional state.

DETAILED DESCRIPTION:
Investigators aims to restore the intestinal bacteria homeostasis through FMT by retention enema with fresh bacteria,thus minimizing bacterial translocation and alleviating infectious complications. The investigators will further examine the effect of FMT on the incidence of infectious complications，duration of clinical course and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of severe acute pancreatitis from the First Affiliated Hospital of Nanchang University according to the Classification of acute pancreatitis-2012: revision of the Atlanta classification and definitions by international consensus
2. Onset of pancreatitis more than 2 weeks
3. Intestinal bacterium screening tips gut dysbacteriosis
4. Patients with symptoms of infection, such as fever, abdominal pain or blood culture and pancreatic necrosis drainage culture positive patients.

Exclusion Criteria:

1. SAP complicated by Gastrointestinal bleeding or Intestinal fistula
2. Pregnancy and lactation women
3. Not signed the informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The control of infectious complications | From admission to discharge
  The temperature recovered to normal for 3 days. The inflammatory cytokines decreased to the normal value.

SECONDARY OUTCOMES:
C-reactive protein（CRP）level | 1day before intervention，7days and 14days after intervention
  C-reactive protein (CRP) is a inflammatory prognostic marker
Procalcitionin（PCT）level | 1day before intervention，7days and 14days after intervention
  Procalcitionin（PCT）level is a inflammatory prognostic marker
Length of Intensive care time and hospital stay | From admission to discharge
  The time of stay in the intensive care unit and hospital
Mortality | From admission to discharge
  The incidence of death during the time frame

CONTACTS AND LOCATIONS:
Overall Officials: Nonghua Lv, MD, Study Chair — the Frist Affiliated Hospital of Nanchang University
Locations (1):
- the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

REFERENCES:
- [Background] Liang J, Sha SM, Wu KC. Role of the intestinal microbiota and fecal transplantation in inflammatory bowel diseases. J Dig Dis. 2014 Dec;15(12):641-6. doi: 10.1111/1751-2980.12211. PMID 25389085
- [Background] Li Q, Wang C, Tang C, He Q, Zhao X, Li N, Li J. Therapeutic modulation and reestablishment of the intestinal microbiota with fecal microbiota transplantation resolves sepsis and diarrhea in a patient. Am J Gastroenterol. 2014 Nov;109(11):1832-4. doi: 10.1038/ajg.2014.299. No abstract available. PMID 25373588
- [Background] Peterson CT, Sharma V, Elmen L, Peterson SN. Immune homeostasis, dysbiosis and therapeutic modulation of the gut microbiota. Clin Exp Immunol. 2015 Mar;179(3):363-77. doi: 10.1111/cei.12474. PMID 25345825
- [Background] Besselink MG, van Santvoort HC, Renooij W, de Smet MB, Boermeester MA, Fischer K, Timmerman HM, Ahmed Ali U, Cirkel GA, Bollen TL, van Ramshorst B, Schaapherder AF, Witteman BJ, Ploeg RJ, van Goor H, van Laarhoven CJ, Tan AC, Brink MA, van der Harst E, Wahab PJ, van Eijck CH, Dejong CH, van Erpecum KJ, Akkermans LM, Gooszen HG; Dutch Acute Pancreatitis Study Group. Intestinal barrier dysfunction in a randomized trial of a specific probiotic composition in acute pancreatitis. Ann Surg. 2009 Nov;250(5):712-9. doi: 10.1097/SLA.0b013e3181bce5bd. PMID 19801929
- [Background] Gu WJ, Liu JC. Probiotics in patients with severe acute pancreatitis. Crit Care. 2014 Jul 3;18(4):446. doi: 10.1186/cc13968. No abstract available. PMID 25043372
- [Background] Cui LH, Wang XH, Peng LH, Yu L, Yang YS. [The effects of early enteral nutrition with addition of probiotics on the prognosis of patients suffering from severe acute pancreatitis]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2013 Apr;25(4):224-8. doi: 10.3760/cma.j.issn.2095-4352.2013.04.011. Chinese. PMID 23660099
- [Background] Tellado JM. Prevention of infection following severe acute pancreatitis. Curr Opin Crit Care. 2007 Aug;13(4):416-20. doi: 10.1097/MCC.0b013e32826388b2. PMID 17599012
- [Background] Hooijmans CR, de Vries RB, Rovers MM, Gooszen HG, Ritskes-Hoitinga M. The effects of probiotic supplementation on experimental acute pancreatitis: a systematic review and meta-analysis. PLoS One. 2012;7(11):e48811. doi: 10.1371/journal.pone.0048811. Epub 2012 Nov 13. PMID 23152810
- [Background] Aroniadis OC, Brandt LJ. Intestinal microbiota and the efficacy of fecal microbiota transplantation in gastrointestinal disease. Gastroenterol Hepatol (N Y). 2014 Apr;10(4):230-7. PMID 24976806
- [Background] Seekatz AM, Aas J, Gessert CE, Rubin TA, Saman DM, Bakken JS, Young VB. Recovery of the gut microbiome following fecal microbiota transplantation. mBio. 2014 Jun 17;5(3):e00893-14. doi: 10.1128/mBio.00893-14. PMID 24939885